CLINICAL TRIAL: NCT01282606
Title: An Open Label, Non-randomized Dose-escalation Study to Assess Safety and Tolerability of SI-6603 in Patients With Lumbar Disc Herniation (Phase II Study)
Brief Title: Clinical Trial to Assess Safety of SI-6603 in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6603/1121
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Vertebra Hernia
Keywords: Chemonucleolysis; Lumbar Vertebrae; Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drug I: SI-6603 (Low) (Experimental)
  Interventions: Drug: SI-6603
- Drug II: SI-6603 (Middle) (Experimental)
  Interventions: Drug: SI-6603
- Drug III: SI-6603 (High) (Experimental)
  Interventions: Drug: SI-6603

INTERVENTIONS:
Drug: SI-6603 — SI-6603 is administrated into the nucleus pulposus of an intervertebral disc.

SUMMARY:
The purpose of this study is to evaluate the safety of SI-6603 in lumbar disc herniation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar disc herniation (L4-L5 or L5-S1) as assessed by MRI and clinical symptoms corresponding to position of the impaired nerve root.
* Patients assessed as positive in the SLR test.
* Patients with sciatica in either lower leg.
* Patients with no improvement from pharmacotherapy or concomitant treatment with drug and nerve block.

Exclusion Criteria:

* Patients who have 2 or more lumbar disc herniations as assessed by MRI.
* Patients with "extrusion-type" or "sequestration-type" herniation in whom a rupture into the posterior longitudinal ligament is identified by MRI.
* Patients who have received nerve block within 3 weeks before screening.
* Patients who have undergone lumbar operation, chemonucleolysis, or percutaneous nucleotomy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | 52 weeks

SECONDARY OUTCOMES:
The leg pain | At each assessment time point

CONTACTS AND LOCATIONS:
Locations (1):
- SKK, Encinitas, California, United States